CLINICAL TRIAL: NCT03437343
Title: Evaluation of Surgeon Performance to Restore Leg Length and Evaluation of the Quality of Life After Total Hip Replacement Related to the Reconstructed Anatomy With EOS Imaging System
Brief Title: Leg Length and Quality of Life After Total Hip Arthroplasty
Acronym: EOS-PTH
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Région Ile de France, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI17039J; 2017-A03333-50 (Registry Identifier: ANSM)
Record Dates: First submitted 2018-02-02; First posted 2018-02-19 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Total Hip Arthroplasty
Keywords: EOS; total hip arthroplasty; performance of surgeons; leg length discrepancy; HOOS
MeSH Terms: conditions — Leg Length Inequality | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Hip arthroplasty

SUMMARY:
This study used 3D reconstructions from the EOS biplanar radiographic imaging system to perform leg length measurements before and after THA (Total hip arthroplasty) on all included THA patients from 2015 to evaluate surgeon performance in restoring lower limb length after THA and the relationships between the quality of life, estimated by the HOOS score (Hip disability and osteoarthritis outcome score), and the anatomy of the new hip in standing position.

DETAILED DESCRIPTION:
The study was conducted in patients who underwent a total hip arthroplasty in Lariboisiere Hospital, Paris, France, during the year 2015.

This retrospective study used 3D reconstructions from the EOS biplanar radiographic imaging system (EOS imaging, Paris, France) to perform leg length measurements before and after THA on all included THA patients from 2015 to evaluate surgeon performance in restoring lower limb length after THA. Included patients either had hip osteoarthritis or femoral head osteonecrosis. Patients were excluded if they were undergoing revision surgery, or had a contralateral THA or total knee.

The performance of the surgeons was judged using the Cumulative Sum control chart (CUSUM) method.

Our objective was to study surgeon performance, measured by their ability to restore the initial preoperative length of the operated leg or to equalize the length of the two legs, and evaluate the relationships between the quality of life, estimated by the HOOS score, and the anatomy of the new hip in standing position using the EOS imaging system.

ELIGIBILITY:
Inclusion Criteria:

* unilateral total hip replacement for osteoarthritis or avascular necrosis healthy contralateral hip
* age over 18 years
* informed consent to participate in the study
* radiographs obtained after total hip replacement using the EOS imaging system, filled HOOS form
* clinical follow-up of 12 months at least

Exclusion Criteria:

* past history of contralateral hip replacement
* ipsi or contralateral knee replacement
* hip arthroplasty performed using a Kerboull cross
* post-operative complications such as infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study was conducted in patients who underwent a total hip arthroplasty in Lariboisiere Hospital, Paris, France, during the year 2015.
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Change in anatomic lower limb length measurements between preoperative and postoperative measurements | preoperative measurements (up to 1 year before surgery) and postoperative measurements (at 1 month after surgery)

SECONDARY OUTCOMES:
Change in flessum/recurvatum/HKS angle (hip knee shaft ) measurements, between preoperative and postoperative measurements | preoperative measurements (up to 1 year before surgery) and postoperative measurements (at 1 month after surgery)
HOOS score (Hip disability and osteoarthritis outcome score) | 24 months after surgery
  The outcome score consists of 40 items assessing 5 subscales. Pain (P) includes 10 items with a total score of 40 points, Symptoms (S) includes 5 items with a total score of 20, Activity limitations daily living (ADL) includes 17 items with a total score of 68 and finally Function in sport and recreation (SP) and hip related quality of life both include 4 items with a total score of 16 each.
  To answer the questions, standardized answer options are given with scores from 0 to 4 (no, mild, moderate, severe and extreme).
  To interpret the score, the outcome measure is transformed in a worst to best scale from 0 to 100, with 100 indicating no symptoms and 0 indicating extreme symptoms.
  To calculate the total HOOS score the subscales need to be summed up, using following formula for all dimension.
  100 - [(patient's score of the subscale x 100)/(total score of the subscale)]